CLINICAL TRIAL: NCT04369885
Title: Assessing Adherence to Home Telemedicine in Individuals With COPD
Brief Title: Assessing Adherence to Home Telemedicine in Individuals With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Midmark Corporation (Industry); Monitored Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-0107
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: home telemedicine; home spirometer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention consisting of a home telemedicine tablet platform (GoHome) that will collect multiple spirometry tests each week (including both forced and slow spirometry measurements), pulse oximetry, and quality of life (QoL) Questionnaire responses. The platform will remind patients to take their medications remind patients to perform measurements, send patients helpful information, and execute a University of North Carolina (UNC) clinic established COPD Action Plan.The backend of the platform is a remote server (Monitored Therapeutics Incorporated CarePortal) that collects the data, send out alerts to the Principal Investigator and can track and trend the data for them.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Home Telemedicine Device (Experimental): This arm will receive the intervention of the home telemedicine device for three months.
  Interventions: Device: Go Home tablet with linked GoSpiro and 3230 Pulse Oximeter

INTERVENTIONS:
Device: Go Home tablet with linked GoSpiro and 3230 Pulse Oximeter — All participants will receive the intervention consisting of a home telemedicine tablet platform (GoHome) that will collect multiple spirometry tests each week (including both forced and slow spirometry measurements), pulse oximetry, and QoL Questionnaire responses. The platform will remind patients to take their medications remind patients to perform measurements, send patients helpful information, and execute a UNC clinic established COPD Action Plan.The backend of the platform is a remote server (Monitored Therapeutics CarePortal) that collects the data, send out alerts to the Principal Investigator and can track and trend the data for them.

SUMMARY:
This is a single-site feasibility pilot study to determine if patients with COPD with an increased risk of exacerbation will use an in-home COPD telemonitoring system for three months that collects lung measures, pulse oximetry, and medication compliance.

DETAILED DESCRIPTION:
This is a single-site, prospective, open label trial evaluating home telemonitoring for patients with COPD and a history of increased exacerbation risk. The purpose of this study is to determine whether automated home monitoring of medication compliance and biometric parameters [forced expiratory capacity in one second (FEV1), forced vital capacity (FVC), peak inspiratory flow rate (PIFR), inspiratory capacity (IC), pulse oximetry, and symptoms] is acceptable to patients, can improve adherence, and may improve clinical outcomes and reduce exacerbations and avoidable 30-day readmissions. Slow spirometry will be performed Sundays, Mondays, Wednesdays, Fridays and Saturdays. Forced spirometry will be performed Tuesdays and Thursdays.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients
* 40 to 80 years of age
* English speaking
* Spirometry confirmed COPD (post-bronchodilator FEV1/FVC<0.70) and post-bronchodilator FEV1% predicted <80% at screening visit. (Target 50% of recruitment with post-bronchodilator FEV1<50% predicted (severe obstruction))
* Increased COPD exacerbation risk defined as either of the following in the prior 12 months:

  * One hospitalization for COPD exacerbation
  * Two outpatient COPD exacerbations requiring treatment with steroids and/or antibiotics
* Signed informed consent

Exclusion Criteria:

* Unable to perform spirometry on their own following training.
* Planned discharge to a nursing home or other extended care facility
* Co-morbid conditions likely to result in non-preventable readmissions (e.g., terminal malignancy, cirrhosis or end-stage liver disease, chronic wound infections, etc.)
* Uncontrolled or untreated medical conditions that would predispose the patient to recurrent COPD exacerbations (i.e., bronchiectasis)
* Patient refusal to or inability to comply with monitoring requirements, for any reason including but not limited to dementia, a history of dementia, or other significant mental impairment
* Patients enrolled in any other clinical trials or therapeutic studies of drugs, devices, or biologics

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Drummond, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Meadowmont Marsico Lung Research Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Home Telemedicine Device
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Home Telemedicine Device
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Home Device Measurement Collection Adherence
Description: Percentage of participants achieving >50% completion of all planned device measurements (spirometry, pulse oximetry and questionnaires) over three months
Time Frame: 3 months
Population: Data were reported for all participants who completed all 3 device component measurements over the entire 3-month study duration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Home Telemedicine Device
Number analyzed (Participants) | 8
percentage of participants | 63 [25 to 91]

2. Primary Outcome: Percentage of Participants With Decrease in COPD Assessment Test (CAT) Score
Description: Percentage of participants achieving ≥2 point decrease in CAT from baseline to three months. The CAT is a short, self-completed, 8-item questionnaire, each item is rated on a 6-point scale ranging from 0 (no impairment) to 5 (maximum impairment). The total CAT score is calculated by summing the scores of all items and ranges from 0 to 40, higher scores indicating severe condition.
Time Frame: 3 months
Population: Data were reported for all participants who completed both initial and final CAT score over the entire 3-month study duration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Home Telemedicine Device
Number analyzed (Participants) | 7
percentage of participants | 57 [18 to 90]

3. Secondary Outcome: Percentage of Participants With Individual Survey Domains Score of 4 or Higher
Description: The percentage of participants with score of 4 or higher on individual survey domains. A satisfaction survey (investigator-developed, 13 questions, each question is graded on a scale of 1-5, 1 being not at all and 5 being extremely) will be used to measure home spirometry and table ease and usefulness.
Time Frame: 3 months
Population: Data were reported for all participants who completed the final survey at the 3-month visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Home Telemedicine Device
Number analyzed (Participants) | 11
percentage of participants
  COPD Prevented Spirometry Use | 36 [11 to 69]
  Spirometer Ease of Use | 46 [17 to 77]
  Spirometer Helpful in Symptom Management | 46 [17 to 77]
  Spirometer Helpful for Identifying Health Problems | 46 [17 to 77]
  Spirometer Helpful for Doctor | 55 [23 to 83]
  Spirometer Helpful for Safety & Security | 73 [39 to 94]
  Willingness to Continue Spirometer Use | 45 [17 to 77]
  Likelihood to Recommend Spirometer | 82 [48 to 98]
  Appeal of Animated Respiratory Therapist Character | 64 [31 to 89]
  Tablet Ease of Use | 82 [48 to 98]
  Tablet Helpful in Symptom Management | 73 [39 to 94]
  Likelihood to Recommend Tablet | 44 [14 to 79]
  Appeal of Tablet | 82 [49 to 98]

4. Secondary Outcome: Median Communication Frequency Survey Score at 3 Months
Description: The median score on a survey question focused on frequency of communication between device and participant. A survey question (investigator-developed, single question) included a scale of 1-5, 1 being "way too much" and 5 being "I wanted a lot more".
Time Frame: 3 months
Population: Data were reported for all participants who completed the final survey at the 3-month visit.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Home Telemedicine Device
Number analyzed (Participants) | 11
score on a scale | 3 [3 to 3]

5. Secondary Outcome: Median Number of Ideal Daily Questions Score at 3 Months
Description: The median score on a survey question focused on the ideal number of questions asked by the device per day. A survey question (investigator-developed, single question) asking participants to indicate how many questions per day was "right" with choices ranging from "1" to "5 or more."
Time Frame: 3 months
Population: Data were reported for all participants who completed the final survey at the 3-month visit.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Home Telemedicine Device
Number analyzed (Participants) | 11
score on a scale | 5 [4 to 5]

6. Secondary Outcome: Rate of Self-reported COPD Exacerbations
Description: The 30-day COPD exacerbation rate, defined as the mean number of events/30 days of follow-up (using three months of follow-up data). COPD exacerbation events are defined as self-reported COPD exacerbations requiring treatment with antibiotics or steroids.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: exacerbations per 30 days
Arm/Group | Home Telemedicine Device
Number analyzed (Participants) | 12
exacerbations per 30 days | 0.14 [0.00 to 0.28]

ADVERSE EVENTS:
Time Frame: From signing of informed consent throughout duration of study, a total of approximately 3 months.
Arm/Group | Home Telemedicine Device
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT04369885/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT04369885/ICF_001.pdf